CLINICAL TRIAL: NCT04953949
Title: First-in-Human Trial of the Safety and Performance of NU-MAX® (IEIK13) as a Hemostatic Agent in Intracranial Neurosurgery
Brief Title: IEIK13 For Neurosurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 3-D Matrix Europe SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEIK13-01
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Oozing (Hemorrhage) During Intracranial Procedures
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Intervention Model Description: Prospective, single arm, multi-center study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NU-MAX® (Experimental): Topical Hemostat
  Interventions: Device: NU-MAX®

INTERVENTIONS:
Device: NU-MAX® — Topical Hemostat

SUMMARY:
The objective of this clinical investigation is to determine the performance and safety profile of NU-MAX® when used as a topical hemostat for oozing bleedings encountered during intracranial procedures, in which control of bleeding by conventional hemostatic techniques is either ineffective or impractical.

ELIGIBILITY:
Inclusion Criteria:

1. Have been informed on the nature of the clinical investigation and provided written informed consent, prior to initiation of any study activities.
2. Able and willing to comply with the clinical investigation follow-up schedule.
3. Male or female human subjects aged 18 years or older at time of enrollment.
4. Requiring hemostasis during elective intracranial procedures, in which the intradural space is accessed and where the control of bleeding by conventional hemostatic techniques is either ineffective or impractical.
5. NU-MAX® is used at least once intraoperatively.

Exclusion Criteria:

1. Patients undergoing emergency craniotomy for traumatic lesions or patients undergoing surgery for primary intracranial hemorrhage.
2. Patients undergoing surgical procedures using a transsphenoidal approach.
3. Intraoperative use of a different topical chemical hemostatic agent prior to the use of NU-MAX® during the same procedure and on the same bleeding point or in the same resection cavity.
4. Patients with a coagulation disorder or medical treatment affecting coagulation or platelet function, unless corrected or stopped prior to surgery.
5. Pregnant patients or patients planning to become pregnant during the clinical investigation.
6. Patients with known allergies to any of the components of NU-MAX®.
7. Patients currently participating in, or having been recently exited from (within 30 days from enrollment in this clinical investigation), or planning to enroll in another clinical investigation that may impact participation or outcomes (at the discretion of the sponsor) of this clinical investigation.
8. Patients with a condition, disorder, or other factor that, in the investigator's opinion, would interfere with study participation.
9. Fever (body temperature >38.5°C) prior to surgery, on the day of the procedure.
10. Patients with a Nickel allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-11-04 (Actual)

PRIMARY OUTCOMES:
% of bleedings reaching hemostasis within 3 minutes | Intraoperatively
  The percentage of bleedings reaching hemostasis within 3 minutes will be measured intraoperatively after the use of NU-MAX® (with a maximum of 3 measurements of hemostasis by NU-MAX® application per subject).

SECONDARY OUTCOMES:
% of bleedings reaching hemostasis within 6 minutes | Intraoperatively
  The percentage of bleedings reaching hemostasis within 6 minutes will be measured intraoperatively after the use of NU-MAX® (up to 3 measurements per subject).

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital (UZA), Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No